CLINICAL TRIAL: NCT04812015
Title: Optimizing Transdiagnostic Non-invasive Vagus Nerve Stimulation to Enhance Learning
Brief Title: Learning and Ear Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00107689
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Learning; taVNS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Dose Group 1 (Other)
  Interventions: Device: transcutaneous auricular vagus nerve stimulation (taVNS) 15 minutes
- Dose Group 2 (Other)
  Interventions: Device: taVNS 30 minutes
- Dose Group 3 (Other)
  Interventions: Device: taVNS 45 minutes
- Dose Group 4 (Other)
  Interventions: Device: taVNS 60 minutes
- Dose Group 5 (Other)
  Interventions: Device: taVNS 75 minutes
- Dose Group 6 (Other)
  Interventions: Device: taVNS 0 minutes

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation (taVNS) 15 minutes — Sham 60 minutes and taVNS active stimulation for 15 minutes
  Arms: Dose Group 1
Device: taVNS 30 minutes — Sham 45 minutes and taVNS active stimulation for 30 minutes
  Arms: Dose Group 2
Device: taVNS 45 minutes — Sham 30 minutes and taVNS active stimulation for 45 minutes
  Arms: Dose Group 3
Device: taVNS 60 minutes — Sham 15 minutes and taVNS active stimulation for 60 minutes
  Arms: Dose Group 4
Device: taVNS 75 minutes — Sham 0 minutes and taVNS active stimulation for 75 minutes
  Arms: Dose Group 5
Device: taVNS 0 minutes — Sham taVNS 75 minutes
  Arms: Dose Group 6

SUMMARY:
This study aims to determine how non-invasive ear stimulation affects learning. During this study, participants will be asked to complete surveys and come to a lab for about 2.5 hours. Researchers will measure brain waves and other body responses (heart rate), while while the ear is stimulated. Participants also will be asked to complete computer tasks. Because brain activity will be measured, participants will be asked to come to the study with clean, dry hair. The study is at MUSC in Charleston. Participants will be compensated for their time. To be eligible, participants must be 18-65 years old, be able to commit 2.5 hours of time to the study, and be able to wear sensors on their hands, arms, and head and sit quietly at a computer.

There are some risks to completing this study. Some questions in the surveys ask about personal thoughts and feelings. The ear stimulation may cause tingling sensations or irritation around the ear.

There are no direct benefits to participants. This study will help researchers improve this ear stimulation as a treatment method.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Non-treatment-seeking community members who do not have a mental health diagnosis and individuals seeking treatment for an anxiety, mood, trauma-related, or obsessive-compulsive disorder.
* Treatment and non-treatment-seeking community members with anxiety, mood, trauma-related, or obsessive-compulsive disorder or symptoms.

Exclusion Criteria:

* Diagnosis of COVID-19 in the past 14 days
* Facial or ear pain or recent ear trauma
* Metal implant devices in the head, heart or neck
* History of brain stimulation or other brain surgery
* History of myocardial infarction or arrhythmia, bradycardia
* Use of B-blockers, antiarrhythmic medication (sodium/potassium/calcium-channel blockers), or blood pressure medications.
* Active respiratory disorder
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury
* Individuals suffering from frequent/severe headaches
* Individuals with lifetime evidence of severe psychiatric disorder (e.g., schizophrenia) or neurological disorder.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5
Started | 6 | 6 | 5 | 6 | 5
Completed | 6 | 6 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 28
Age, Categorical [Count of Participants; unit: Participants] — Date of Birth and Reported continuous age
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 6 | 6 | 5 | 6 | 5 | 28
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (8.4) | 34.5 (12.3) | 38.2 (16.9) | 32.7 (15.9) | 26.8 (3.0) | 32.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Dose 1- 1 participant declined to report their sex
  Participants
    number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 27
    Female | 3 | 4 | 3 | 4 | 3 | 17
    Male | 2 | 2 | 2 | 2 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 4 | 6 | 5 | 24
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 5 | 6 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in P300 Amplitude
Description: Measured for standard versus deviant tones during the Auditory Oddball Task. Oddball will be administered at 2 intervals during stimulation.
Time Frame: Measured at Baseline and last 10 minutes of stimulation, on average 65 minutes
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 5
microvolts | .88 (2.01) | .50 (1.4) | -.15 (1.8) | -.26 (.61) | .23 (1.4)

2. Primary Outcome: Change in Heart Rate Variability
Time Frame: Baseline to end of Active Stimulation
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 4
ms | 2.9 (1.6) | 1.9 (.7) | 1.5 (1.1) | 1.3 (.2) | 1.7 (.6)

ADVERSE EVENTS:
Time Frame: 1 Day
Description: Definitions of adverse event and serious adverse event are similar to clinicaltrials.gov.
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT04812015/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04812015/ICF_001.pdf